CLINICAL TRIAL: NCT06422585
Title: Comparison of Three Different Analgesic Nerve Blocks in Total Knee Replacement Surgery
Brief Title: Comparison of Different Analgesic Nerve Blocks in Total Knee Replacement Surgery
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Serena Ricalzone, principal investigator, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: PGBLOCK
Record Dates: First submitted 2024-04-26; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Knee Prosthesis; Pain, Procedural
Keywords: Knee; Post procedural pain; Regional anesthesia
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Femoral Nerve Block + IPACK Block: After adequate venous access has been obtained, spinal anesthesia with Levobupivacaine will be performed. After which antalgic Femoral Nerve Block and IPACK Block will be performed.
- Saphenous (Adductor Canal) Block + IPACK Block: After adequate venous access has been obtained, spinal anesthesia with Levobupivacaine will be performed. After which Saphenous and IPACK Block will be performed.
- Dual Subsartorial Block: After adequate venous access has been obtained, spinal anesthesia with Levobupivacaine will be performed. After which Dual Subsartorial Block will be performed.

SUMMARY:
The goal of this observational study is to compare the equivalent analgesic efficacy of three regional anesthesia techniques in total knee replacement surgery. The main question it aims to answer is:

• Non inferiority of each technique in relation to the others Participants will receive selective spinal anesthesia and the antalgic nerve block depending on the group they happen to be in.

Researchers will compare the Femoral Nerve Group+IPACK block, the Saphenous Nerve block+IPACK and the Subsartorial Block groups to see if there is any difference in the pain control in the 24 hours after the surgery.

DETAILED DESCRIPTION:
After adequate venous access is obtained, a light sedation with Midazolam 1-2 mg is administered. The patient will be monitored and a selective spinal anesthesia will be performed. After the neuraxial procedure the antalgic block of choice is performed with about 40 mL of long acting local anesthetic.

Magnesium Solfate 1g and Dexametasone 4mg are administered after the block. If the patient wishes, a propofol continuos infusion may be administered for sedation during the surgery. Before the patient leaves the OR, Ketorolac 30mg will be administered.

Pain control after surgery will be achieved with acetaminophen 1g t.i.d., Ketorolac 30mg on demand, and Morphine solfate if NRS >5 after Ketorolac.

Every 6 hours the patient will be monitored by the anesthesia team. After 24 hours the antalgic effect of the nerve block is reasonably thought to be over, so the follow up is interrupted.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y/o
* Total knee replacement elective surgery
* Informed consent

Exclusion Criteria:

* Age < 18 y/o
* Surgery with general anesthesia
* Patients with coagulopaties
* Patients in chronic opioid therapy
* Refuse to sign informed consent form
* Unable to sign informed consent form
* Know allergies to medication used for analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
NRS | Baseline, every 6 hours for the first 24 hours after surgery
  To compare the analgesic effect at 24 hours, of a nerve block technique compared to others after selective spinal anesthetic is administerd to achieve surgical anesthesia.Evaluate pain for every group in the first 24 hours post surgery using the Numeric Pain Scale (NRS) assigning a numeric value between zero (no pain) and ten (the worst pain ever felt). Absence of relevant pain is considered a NRS less than three.
  Success of the block was defined as NRS≤3.

SECONDARY OUTCOMES:
side effect | 24 hours
  Monitoring the onset of side effects (nausea/vomiting/hypotension/dizziness/sensitive impareiment) in every group of patients in the first 24 hours every six hours

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Nardi, MD, Study Director — Azienda Ospedaliera Universitaria Pisana; Alessandro Cardu, MD, Study Chair — Scuola Specializzazione - Università di Pisa
Locations (1):
- Edificio 3 - Azienda Ospedaliero Universitaria Pisana Cisanello, Pisa, Tuscany, Italy